CLINICAL TRIAL: NCT00699322
Title: The Comparative Study of Dipeptidyl Peptidase-IV Inhibitor and Sulfonylurea on the Effect of Improving Glucose Variability and Oxidative Stress in Type 2 Diabetic Patients With Inadequate Glycemic Control on Metformin
Brief Title: Effect of Dipeptidyl Peptidase-IV Inhibitor and Sulfonylurea on Glucose Variability and Oxidative Stress
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Collaborators: MSD Korea Ltd. (Industry)
Responsible Party: Kun-Ho Yoon, Kangnam St.Mary's hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCMC08MI081
Record Dates: First submitted 2008-06-16; First posted 2008-06-17 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Type 2 Diabetes
Keywords: glucose variability; oxidative stress; sitagliptin; glimepiride
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Sitagliptin
  Interventions: Drug: Sitagliptin
- 2 (Active Comparator): Glimepiride
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Sitagliptin — 100mg P.O. per day for 1month
  Other Names: Januvia
  Arms: 1
Drug: Glimepiride — 2mg P.O. per day for 1 month
  Other Names: Glimel
  Arms: 2

SUMMARY:
This research will focus on the effect of Sitagliptin on 24 hour glycemic excursion and improvement of oxidative stress markers compared to long acting sulphonylurea Glimepiride in type 2 diabetic patients with inadequate glycemic control on metformin

DETAILED DESCRIPTION:
Sitagliptin might improve not only the mean glycemic control during study period but also 24 hour glycemic fluctuation by restoring the physiologic pattern of insulin secretion. Furthermore decrease postprandial glycemic excursion should decrease the oxidative stress markers. Those effects might be amplified in Asian patients because of prominent early phase insulin secretory defects accompanied with relatively less degree of insulin resistance. Based on this assumption, this research will focus on the effect of Sitagliptin on 24 hour glycemic excursion and improvement of oxidative stress markers compared to long acting sulphonylurea Glimepiride in type 2 diabetic patients with inadequate glycemic control on metformin.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes
* duration of diabetes less than 10 years
* HbA1c 6.5-8.0%
* BMI 20-30
* on stable dose of metformin (more than 1000mg) for at least 2 months

Exclusion Criteria:

* having oral hypoglycemic agents other than metformin
* using insulin
* serum creatinin >= 1.5 mg/dL
* SGOT, SGPT >= 90
* ischemic heart disease
* congestive heart failure (NYHA class >=2)
* severe diabetic complication (PDR, CRF, CVA)
* on medication affecting glucose profile (such as steroid)
* infectious disease
* malignancy
* pregnant or breast-feeding woman

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Glucose variability | 1 month

SECONDARY OUTCOMES:
oxidative stress markers (oxidized LDL, N-carboxymethyl-lysine(CML), nitrotyrosine, 8-iso-prostaglandinF2α, 8-OhDG) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ho Yoon, M.D., Ph.D., Principal Investigator — Kangnam St.Mary's hospital
Locations (1):
- Kangnam St. Mary's hospital, Seoul, South Korea

REFERENCES:
- [Background] Monnier L, Mas E, Ginet C, Michel F, Villon L, Cristol JP, Colette C. Activation of oxidative stress by acute glucose fluctuations compared with sustained chronic hyperglycemia in patients with type 2 diabetes. JAMA. 2006 Apr 12;295(14):1681-7. doi: 10.1001/jama.295.14.1681. PMID 16609090
- [Background] Colette C, Monnier L. Acute glucose fluctuations and chronic sustained hyperglycemia as risk factors for cardiovascular diseases in patients with type 2 diabetes. Horm Metab Res. 2007 Sep;39(9):683-6. doi: 10.1055/s-2007-985157. PMID 17846977